CLINICAL TRIAL: NCT05622175
Title: A Dose-finding Phase I Study of F8IL10 Intra-articular Treatment in Rheumatoid Arthritis
Brief Title: Safety and Preliminary Signs of Efficacy of F8IL10 for Intra-articular Treatment
Acronym: DekaJoint
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study redesigned and registered under NCT07245992 (Protocol n° PH-F8IL10INTRA-03/24)
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH-F8IL10INTRA-02/22
Record Dates: First submitted 2022-11-03; First posted 2022-11-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: Dose escalation of F8IL10 to determine the MTD and the RD when administered intra-articular. A standard 3+3 dose escalation design from 0.5 to 10 mg of F8IL10 until the first instance of a DLT in the observation period from Day 1 to Day 28. In the absence of DLTs, such dose increase will continue until the MAD level is reached and won't exceed 10 mg dose level. With the occurrence of a DLT, the same dose level cohort will be expanded to 6 patients and, if additional DLTs do not occur, the dose escalation will continue to the next dose level. When two DLTs are recorded in the same dose level, MAD is automatically reached. The RD will be then defined by the DSMB .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drug: F8IL10 (Experimental): Overall, 32 patients will participate in case no DLT would occur.
  1. In the standard 3+3 dose escalation part, participants will be enrolled in cohorts and will be treated with different doses of F8IL10 (from 0.5 to 10 mg) in order to identify a RD to be further explored in the subsequent dose expansion part. In the dose escalation part, patients will be treated in cohorts of 3 patients with escalating doses of F8IL10 until the MAD is reached and won't exceed 10 mg dose level. In case a DLT would be detected, further 3 patients will be enrolled for that cohort in order to confirm the MAD or to proceed with the next dose level. Therefore, up to 30 patients could be enrolled in the dose escalation part.
  2. Following successful identification of the RD, the study will proceed with a dose expansion part and 20 patients will be treated at the RD dose level (patients treated at the RD in the course of the dose escalation phase will contribute to the total sample size).
  Interventions: Drug: F8IL10

INTERVENTIONS:
Drug: F8IL10 — The study consists of a dose escalation of F8IL10 to determine the MTD and the RD when administered intra-articular.
  Patients with arthritis flare(s) in "large joints" (shoulders, elbows, knees and ankles, with the exception of hip) and "small joints" (metacarpophalangeal joints, proximal interphalangeal joints, second through fifth metatarsal-phalangeal joints, thumb interphalangeal joints, and wrists) defined as per "2010 Rheumatoid Arthritis Classification Criteria" [1] will be treated with increasing dose of F8IL10 according to the schedule detailed below:
  Cohort 1: 0.5 mg F8IL10 Cohort 2: 1 mg F8IL10 Cohort 3: 2.5 mg F8IL10 Cohort 4: 5 mg F8IL10 Cohort 5: 10 mg F8IL10
  Other Names: Dekavil

SUMMARY:
This multicenter, prospective Phase I study is aimed at testing the safety of F8IL10 via i.a. administration once every 4 weeks over 8 weeks in patients with RA who, despite treatment with stable doses (at least 3 months) of DMARDs (conventional, biologic and/or targeted synthetic), present arthritis flare(s) suitable for i.a. injections.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 and ≤ 80 years.
2. Diagnosis of RA according to ACR/EULAR classification criteria (2010) with a disease duration exceeding 6 months.
3. Presence of at least an arthritis flare suitable for i.a. injection despite treatment with stable doses (for at least 3 months) of DMARDs (conventional, biologic and targeted synthetic) background therapy.
4. Stable regimens of NSAIDs and/or oral corticosteroid (≤ 10 mg/day; prednisone equivalent) for a period ≥ 2 weeks prior to screening.
5. All acute toxic effects of any prior therapy must have returned to classification "mild" according to CTCAE v.5.0 (published on November 27, 2017).
6. Sufficient hematologic, liver and renal function:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥100 x109/L, haemoglobin (Hb) ≥ 10.0 g/dL.
   * Alkaline phosphatase (AP), alanine aminotransferase (ALT) and or aspartate aminotransferase (AST) ≤ 3 x upper limit of normal range (ULN), and total bilirubin ≤ 2.0 mg/dl (34.2 µmol/L).
   * Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 50 mL/min.
7. Documented negative TB test (e.g. Quantiferon or equivalent) and Chest X-ray. Results of tests carried out prior to the participation in the study may be accepted, if deemed as appropriate to exclude active TB by the study physician.
8. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no ongoing infection are eligible. Results of tests carried out prior to the participation in the study may be accepted, if deemed as appropriate to exclude active infections by the study physician.
9. Sexually active male or female patients of childbearing potential are eligible providing that:

   Female:
   * Women of childbearing potential (WOCBP) have a negative pregnancy test performed within 14 days prior to treatment start.
   * WOCBP agree to use, from the screening to 6 months following the last study drug administration, effective method of birth control as applicable per local law that both results in a Pearl index < 1 and considered highly effective as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the "Clinical Trial Facilitation Group" (e.g. combined estrogen and progestogen containing hormonal contraception, progestogen-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, vasectomized partner, total sexual abstinence or bilateral tubal occlusion).

   Male:

   - Agree to use two acceptable methods of contraception (e.g. condom with spermicidal gel) from the screening to 6 months following the last study drug administration. Females of childbearing potential that are partners of male study participants must observe the same birth control indications that apply to female participants.
10. Signed and dated Ethics Committee-approved informed consent form indicating that the patient has been informed of all pertinent aspects of the study.
11. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

Patients must not be enrolled into the study if, at the time of enrollment, they have any of the following:

1. Presence of active infections or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or would interfere with the study objectives or conduct.
2. Pregnancy, lactation or unwillingness to use adequate contraceptive methods.
3. Diagnosis of any other inflammatory arthritis or active autoimmune diseases other than RA.
4. Received intra-articular administration of corticosteroids/DMARDs (for other reasons than the current study) within 4 weeks or 5 half-lives prior to the first dose of study drug, whichever is longer.
5. History or currently active primary or secondary immunodeficiency.
6. Concurrent malignancy or history of malignancy (except in situ melanoma) from which the patient has been disease-free for less than 2 years.
7. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
8. Treatment with warfarin or other coumarin derivatives.
9. Clinically significant cardiac arrhythmias or requiring permanent medication.
10. Abnormal LVEF or any other abnormalities observed during baseline ECG and echocardiogram investigations that are considered as clinically significant by the investigator; subjects with current or a history of QT/QTc prolongation.
11. Uncontrolled hypertension.
12. Known arterial aneurism at high risk of rupture.
13. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche-Fontaine classification).
14. Severe diabetic retinopathy.
15. Major trauma including surgery within 4 weeks prior to administration of study treatment.
16. Known history of allergy or other intolerance to IL10 or other drugs based on human proteins/peptides/antibodies.
17. Treatment with any investigational agent within 4 weeks or 5 half-lives prior to the first dose of study drug, whichever is longer.
18. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline or plan to receive vaccines during the study.
19. Chronic pain disorders (not RA-related) that might interfere with pain evaluation.
20. Patients requiring stable doses of corticosteroids > 10 mg/day (prednisone equivalent). Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
21. History of alcohol, drug or chemical substance abuse within the 6 months prior to screening.
22. Any condition that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MTD | From the enrollment of each patient until the completion of the treatment (for a maximum of 9 weeks)
  Maximum Tolerated Dose (in dose escalation part). The MAD is defined when at least two patients within a cohort of 2-6 patients experience a DLT (i.e., ≥33% of patients with a DLT at that dose level.
RD | From the enrollment of each patient until the completion of the treatment (for a maximum of 9 weeks)
  Recommended Dose (in dose escalation part). The RD is defined by the Data Safety Monitoring Board (DSMB) among the safely tested dose level (i.e. not exceeding the MTD) considering the overall results dataset (e.g. safety, tolerability, efficacy, immunogenicity, pharmacokinetics) obtained in this study.

SECONDARY OUTCOMES:
Safety and Tolerability | From the start of treatment period (for a maximum of 9 weeks) to the end of follow-up period (for a maximum of 6 months)
  Number and frequency of Adverse Events (AEs), Serious Adverse Events (SAEs), Dose Limiting Toxicities (DLTs) and Drug-Induced Liver Injuries (DILIs)
Efficacy measured as improvement in visual analogue scale for involved joint pain (jVAS) | From the start of treatment period (for a maximum of 9 weeks) to the end of follow-up period (for a maximum of 6 months)
  Preliminary efficay findings using jVAS scale in rheumatoid arthritis for quantifying pain intensity. Patients will assess their own current level of pain related to arthritis in target joint(s) that has been/will be injected. The information refers to a score of the joint pain perceived by the patient over the 7 days prior to the assessment and will be recorded using a 100-mm horizontal VAS where the left end represents "no pain (0%)" and the right end represents "severe pain (100%)". The assessment provided at Day 1 (Week 1) will be considered as baseline measurement.
Quality of life - Collection of HAQ-DI for the evaluation of physical function | At day 1 and 29 (F8IL10 administration) to the end of follow-up period (for a maximum of 6 months)
  Health Assessment Questionnaire-Disability Index (HAQ-DI) as validated tool for the evaluation of Disability Index (DI) or Functional Disability Index (FDI) by considering 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 (without any difficulty) to 3 (unable to do). For each section, the score given to that section is the worst score within the section. The 8 scores of the 8 sections are summed and divided by 8. Changes from baseline through treatment period and follow-up will be quantified.
Quality of life - Collection of SF-36 for the evaluation of overall health status | At day 1 and 29 (F8IL10 administration) to the end of follow-up period (for a maximum of 6 months)
  Short Form Health Survey 36 (SF-36) as validated tool for subject-reported indication of overall health status, including multi-item scales measuring 8 health concepts: (1) physical functioning; (2) role limitations because of physical health problems; (3) bodily pain; (4) social functioning; (5) general mental health; (6) role limitations because of emotional problems; (7) vitality; and (8) general health perceptions. These are summarized in two summary measures of physical and mental health: the Physical Component Summary and Mental Component Summary. Lower scores equate to higher disability and higher scores equate to lower disability. Changes from baseline through treatment period and follow-up will be quantified.
Quality of life - Collection of FACIT-F for the evaluation of self-reported fatigue and its impact upon daily activities and function | At day 1 and 29 (F8IL10 administration) to the end of follow-up period (for a maximum of 6 months)
  Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) as validated 13-item questionnaire for the assessment of self-reported fatigue and its impact upon daily activities and function. It uses a 5-point Likert-type scale (0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). As each of the 13 items of the FACIT-Fatigue scale ranges from 0-4, the range of possible scores is 0-52, with 0 being the worst possible score and 52 the best. Changes from baseline through treatment period and follow-up will be quantified.
Assessment of joint inflammation with ultrasound | At day 1 and 57 of treatment period
  Assessment of improvement of joint synovitis using ultrasound (US) pre-treatment and after the treatment period
Assessment of damage with ultrasound | At day 1 and 57 of treatment period
  Assessment of non-progressive bone erosion using ultrasound (US) pre-treatment and after the treatment period
Pharmacokinetic (PK) profile F8IL10- Area Under the Curve (AUC) | At day 1 and 29 (F8IL10 administration)
  Blood/Synovial fluid samples for PK profile of F8IL10 profile measurements will be collected from all patients enrolled in the study and who receives at least one dose of study drug and have adequate PK sampling.
  Standard PK parameter AUC will be estimated.
Pharmacokinetic (PK) profile F8IL10- Maximum drug concentration (Cmax) | At day 1 and 29 (F8IL10 administration)
  Blood/Synovial fluid samples for PK profile of F8IL10 profile measurements will be collected from all patients enrolled in the study and who receives at least one dose of study drug and have adequate PK sampling.
  Standard PK parameter Cmax will be estimated.
Pharmacokinetic (PK) profile F8IL10 - Terminal half-life (T½) | At day 1 and 29 (F8IL10 administration)
  Blood/Synovial fluid samples for PK profile of F8IL10 profile measurements will be collected from all patients enrolled in the study and who receives at least one dose of study drug and have adequate PK sampling.
  Standard PK parameter T½ will be estimated.
Immunogenicity of F8IL10 (Human Anti-Fusion Antibody formation [HAFA]) | At day 1 and 29 (F8IL10 administration) to the first visit of follow up (week 13)
  Blood samples to assess the potential development of antibody formation to F8IL10 will be collected during the treatment period and in the first Follow-up